CLINICAL TRIAL: NCT03044860
Title: Enteroendocrine Cells in Healthy Individuals and Patients With Type 2 Diabetes
Brief Title: Anatomical and Physiological Characterisation of the Gut Endocrine Cells in Healthy and in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, MD, PhD, professor, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Endocrinemapping
Record Dates: First submitted 2017-01-10; First posted 2017-02-07 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type 2 diabetes (Experimental): Adult patients with type 2 diabetes undergoing double-balloon enteroscopy (DBE) with biopsy retrieval using a DBE-device.
  Interventions: Procedure: Double-balloon enteroscopy (DBE) with biopsy retrieval
- Healthy (Experimental): Adult subjects without type 2 diabetes undergoing double-balloon enteroscopy (DBE) with biopsy retrieval using a DBE-device.
  Interventions: Procedure: Double-balloon enteroscopy (DBE) with biopsy retrieval

INTERVENTIONS:
Procedure: Double-balloon enteroscopy (DBE) with biopsy retrieval — With the use of a double-balloon enteroscopy device, study participants underwent upper and lower enteroscopies with mucosal biopsy mucosal biopsy retrieval from every ~30 cm of the small intestine and specific locations in the large intestine

SUMMARY:
Investigation of the anatomical distribution of enteroendocrine cells by a systematic approach along the entire human intestinal tract in healthy individuals and patients with type 2 diabetes.

DETAILED DESCRIPTION:
Enteroendocrine K and L cells are pivotal in regulating appetite and glucose homeostasis, but knowledge of their distribution in man is sparse and it is unknown whether alterations occur in type 2 diabetes. Twelve patients with type 2 diabetes and 12 age and BMI-matched healthy individuals underwent upper and lower double-balloon enteroscopy with mucosal biopsy retrieval from every ~30 cm of the small intestine and specific locations in the large intestine. The investigators evaluated the distribution of enteroendocrine cells (using IHC staining for their specific hormonal products) and evaluated mRNA expression of the corresponding genes along the entire intestinal tract in patients with type 2 diabetes and in healthy individuals.

ELIGIBILITY:
Inclusion criteria:

Type 2 diabetes patients

* Diagnosis of type 2 diabetes (at least 3 months prior to study inclusion)
* Treatment with diet counseling alone or combined with an glucose-lowering drugs: metformin or sulphonylurea
* Caucasian ethnicity
* Age >25 and <70 years
* Normal hemoglobin
* Negative for autoantibodies to glutamic acid decarboxylase (GAD-65) and islet cell autoantibodies (ICA).

Healthy individuals

* Fasting plasma glucose <6.0 mM
* Plasma glucose 2 hours after a 75 g-oral glucose tolerance test <7.8 mM
* Negative for GAD-65 antibodies and ICA
* Caucasian ethnicity
* Age >25 and <70 years
* Normal hemoglobin

Exclusion criteria:

Type 2 diabetes patients

* Liver disease (evaluated by alanine aminotransferase and/or aspartate aminotransferase >2 times normal value)
* Treatment with dipeptidyl peptidase 4 inhibitors or medicine that could not be paused for 12 hours
* Previous hysterectomy, appendectomy, cholecystectomy or caesarean
* Sleep apnea
* American Society of Anesthesiologists class >3
* Allergy to soy protein or eggs
* BMI >35 kg/m2 or any other condition that would contraindicate propofol sedation or enteroscopy.

Healthy individuals

* Liver disease (evaluated by alanine aminotransferase and/or aspartate aminotransferase >2 times normal value)
* Liver disease (evaluated by alanine aminotransferase and/or aspartate aminotransferase >2 times normal value)
* Treatment with dipeptidyl peptidase 4 inhibitors or medicine that could not be paused for 12 hours
* Previous hysterectomy, appendectomy, cholecystectomy or caesarean
* Sleep apnea
* American Society of Anesthesiologists class >3
* Allergy to soy protein or eggs
* BMI >35 kg/m2 or any other condition that would contraindicate propofol sedation or enteroscopy
* First-degree relative(s) with type 1 or type 2 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of enteroendocrine cells (density and mRNA expression) in the intestinal tract. | Cross-sectional study. Each participant went through two study days (upper and lower double-ballon enteroscopy, respectively)
  Using a double-balloon enteroscopy device, mucosal biopsies are obtained from the entire intestinal tract in 12 healthy individuals and 12 patients diagnosed with type 2 diabetes. The biopsies are analysed using immunohistochemistry (IHC) and mRNA expression analysis.
  Positively stained enteroendocrine cells (from IHC) are counted and divided by the epithelial area providing 'density' (cells/mm2).
  The data obtained from cell count and mRNA expression analysis present the variation in number of enteroendocrine cells (density) and the expression of hormonal products along the intestinal tract.
Evaluation of differences in enteroendocrine cells (density and mRNA expression) along the intestinal tract of healthy individuals compared with type 2 diabetes patients. | Cross-sectional study. Each participant went through two study days (upper and lower double-ballon enteroscopy, respectively)
  Using a double-balloon enteroscopy device, mucosal biopsies are obtained from the entire intestinal tract in 12 healthy individuals and 12 patients diagnosed with type 2 diabetes. The biopsies are analysed using immunohistochemistry (IHC) and mRNA expression analysis.
  Positively stained enteroendocrine cells (from IHC) are counted and divided by the epithelial area providing 'density' (cells/mm2).
  Cell count (density) and mRNA expression data obtained from the healthy individuals and type 2 diabetes patietns are compared to evaluate potential differences between the two groups.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gilliam-Vigh H, Ellegaard AM, Madsen MR, Lund AB, Jensen BAH, Vilsboll T, Rigbolt K, Knop FK. Mucosal transcriptomic landscape along the small and large intestines in individuals with and without type 2 diabetes. Gut. 2025 Dec 5;75(1):33-45. doi: 10.1136/gutjnl-2024-334124. PMID 40803750
- [Derived] Gilliam-Vigh H, Suppli MP, Heimburger SMN, Lund AB, Knop FK, Ellegaard AM. Cholesin mRNA Expression in Human Intestinal, Liver, and Adipose Tissues. Nutrients. 2025 Feb 8;17(4):619. doi: 10.3390/nu17040619. PMID 40004948
- [Derived] Gilliam-Vigh H, Jorsal T, Nielsen SW, Forman JL, Pedersen J, Poulsen SS, Vilsboll T, Knop FK. Expression of Secretin and its Receptor Along the Intestinal Tract in Type 2 Diabetes Patients and Healthy Controls. J Clin Endocrinol Metab. 2023 Nov 17;108(12):e1597-e1602. doi: 10.1210/clinem/dgad372. PMID 37335970
- [Derived] Gilliam-Vigh H, Jorsal T, Rehfeld JF, Pedersen J, Poulsen SS, Vilsboll T, Knop FK. Expression of Cholecystokinin and its Receptors in the Intestinal Tract of Type 2 Diabetes Patients and Healthy Controls. J Clin Endocrinol Metab. 2021 Jul 13;106(8):2164-2170. doi: 10.1210/clinem/dgab367. PMID 34036343
- [Derived] Jorsal T, Rhee NA, Pedersen J, Wahlgren CD, Mortensen B, Jepsen SL, Jelsing J, Dalboge LS, Vilmann P, Hassan H, Hendel JW, Poulsen SS, Holst JJ, Vilsboll T, Knop FK. Enteroendocrine K and L cells in healthy and type 2 diabetic individuals. Diabetologia. 2018 Feb;61(2):284-294. doi: 10.1007/s00125-017-4450-9. Epub 2017 Sep 28. PMID 28956082